CLINICAL TRIAL: NCT04114084
Title: Sleep Apnea in Patients With MGUS and MM
Status: Recruiting | Type: Observational
Sponsor: Michael Tomasson (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Michael Tomasson, Professor of Internal Medicine, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202208637-A
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance
MeSH Terms: conditions — Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole exome, genome wide and RNA sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A. patients with MGUS and sleep apnea
  Interventions: Procedure: Bone Marrow Aspirate and Biopsy
- B. patients with MGUS and no sleep apnea
  Interventions: Procedure: Bone Marrow Aspirate and Biopsy
- C. patients with MM and sleep apnea
  Interventions: Procedure: Bone Marrow Aspirate and Biopsy
- D. patients with MM and no sleep apnea
  Interventions: Procedure: Bone Marrow Aspirate and Biopsy

INTERVENTIONS:
Procedure: Bone Marrow Aspirate and Biopsy — The aspirate sample obtained for research at the time a standard-of-care biopsy is taking place will be approximately 40cc. Bone marrow aspiration removes bone marrow fluid and cells through a needle placed into the bone. Usually this sample is taken from the back of the pelvic bone, but it may also be taken from the sternum or the front of the pelvic bone. A bone marrow biopsy removes bone with the marrow inside and is done prior to the aspirate. Each biopsy and aspirate procedure takes approximately 15 minutes total. Bone marrow aspirate may be collected in a separate tube for research or collected from the standard-of-care specimen with left-over aspirate not otherwise needed for clinical purposes, or from previous procedures.

SUMMARY:
This study involves patients with plasma cell dyscrasia including monoclonal gammopathy of undetermined significance (MGUS) or multiple myeloma (MM), with and without sleep apnea, who are providing bone marrow specimens. Specimens will be obtained at the time that patients undergo a standard-of-care procedure in order to minimize discomfort and reduce any risk.

DETAILED DESCRIPTION:
Obesity is a risk factor for the development of MM, although the mechanisms that link obesity and MM are unclear. Obesity, in turn, is closely associated with obstructive sleep apnea. Interestingly, the key risk factors for both sleep apnea and MM are overlapping (age, sex, race and body mass index). During the apnea, or cessation of normal breathing, arterial oxygen saturation falls. This can occur as often as 60 times per hour, resulting in chronic intermittent hypoxia (CIH). In preliminary studies, investigators exposed C57BL/6 mice, that are typically resistant to engraftment of malignant plasma cells to CIH, followed by injection of malignant 5TGM1 cells. With CIH, 5TGM1 cells homed to bone marrow, and engrafted and expanded, resulting in lethal disease. These mice had key features of the myeloma phenotype, including bone damage and gammopathy. Investigators explored potential mechanisms by which CIH promote MM progression by performing whole bone marrow RNASeq analysis. They found pathways relevant to angiogenesis, cell adhesion, and stromal cell development (including dendritic cells and eosinophils) to be upregulated. This is an exciting and potentially translational finding because these elements are also upregulated in the bone marrow of human myeloma patients. Investigators also found upregulation of B cell and plasma cell development and differentiation pathway, and downregulation of B-cell apoptosis pathways. Taking these preliminary findings together, the overarching hypothesis is that CIH increases oxidative stress, thereby supporting B cell maturation and changing the bone marrow stromal microenvironment to drive the progression to MM.

ELIGIBILITY:
Patients diagnosed with MGUS or MM who will be receiving a bone marrow biopsy as part of their standard of care are eligible to participate in this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with MGUS or MM who will be receiving a bone marrow biopsy as part of their standard of care with and without sleep apnea
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2030-05-23 (Estimated); Study Completion 2030-05-23 (Estimated)

PRIMARY OUTCOMES:
To quantify the incidence of sleep apnea and sleep disorder in patients with MGUS and MM | From study initiation up to 5 years
To compare gene expression in bone marrow stroma of MGUS and MM patients, with and without sleep apnea, and following sleep apnea treatment. | From study initiation up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tomasson, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No